CLINICAL TRIAL: NCT00583752
Title: Phase II Study of Adenovirus/PSA Vaccine in Men With Recurrent Prostate Cancer After Local Therapy
Brief Title: Phase II Study of Adenovirus/PSA Vaccine in Men With Recurrent Prostate Cancer After Local Therapy APP21
Acronym: APP21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David M Lubaroff (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David M Lubaroff, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201705743; 200605706 (Other: Initial UI IRB ID number)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Recurrent Prostate Cancer
Keywords: prostate cancer; vaccine; immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Androgen deprivation therapy (ADT) + Adenovirus/PSA Vaccine (Experimental): On Arm B, subjects will be started on androgen deprivation therapy (ADT) 14 days prior to beginning the vaccinations.
  Interventions: Biological: Adenovirus/PSA Vaccine
- Adenovirus/PSA Vaccine (Experimental): On Arm A, subjects can begin the three vaccinations immediately.
  Interventions: Biological: Adenovirus/PSA Vaccine

INTERVENTIONS:
Biological: Adenovirus/PSA Vaccine — 1x10E8pfu in Gelfoam subcutaneously on day 0, 30, 60

SUMMARY:
The purpose of this study is to determine whether vaccination with the Ad/PSA vaccine will induce an anti-PSA immunity that will result in the destruction of the remaining prostate cancer cells.

DETAILED DESCRIPTION:
Subjects will be randomized to Arm A (vaccine only) or Arm B (androgen deprivation therapy plus vaccine). On Arm A, subjects can begin the three vaccinations immediately. On Arm B, subjects will be started on androgen deprivation therapy (ADT) 14 days prior to beginning the vaccinations.

Subjects will be vaccinated three times, each injection administered at 30-day intervals. Based upon our earlier clinical trial, the vaccine is considered safe and should not induce any major side effects. The investigators hope that vaccination with this PSA virus will cause the body to produce immunity to the PSA and that immunity will destroy any cell that produces PSA. Since the only cells left in the body that produce PSA will be the cancer cells, the investigators propose that the vaccination and ensuing anti-PSA immunity will kill the prostate cancer cells. Importantly, this treatment should not cause any major side effects as would treatment with anti-cancer drugs.

ELIGIBILITY:
Inclusion Criteria:

* Men with prostate cancer who have received prior local therapy (radical prostatectomy or definitive radiation therapy) and have biochemical (PSA) relapse without evidence of radiographic or clinical metastatic disease.
* For men who had prior prostatectomy, the surgery must have occurred at least 6 months prior to initiation of treatment.
* For men who had prior definitive radiation therapy, radiation must have been completed at least 1 year prior to initiation of treatment.
* Exhibit at least three separate rises in serum PSA, at least one month apart with differences >/= 0.03 ng/ml and a total PSA of >0.2 ng/ml.
* Have a PSA doubling time of >/= 6 months if the baseline serum PSA was >2 ng/ml.
* Negative bone scans.
* Negative CT scans of abdomen and pelvis (no evidence of soft tissue lesions >/= 1 cm).
* Scans must be obtained within 6 weeks of entry into the trial (initiation of treatment).
* Written informed consent.
* Age >/= 18 years.
* Required laboratory values [obtained within 2 weeks of study entry (initiation of treatment)].
* Serum creatinine </= 2.0 mg/dL
* Adequate hematologic function: granulocytes >/= 1800 per mm3, platelets >/= 100,000 per mm3, WBC >/= 3700, and lymphocytes >/= 590.
* Adequate hepatocellular function: AST <3x upper limit of normal and bilirubin <1.5 mg/dl (unless bilirubin elevation is consistent with Gilbert's syndrome).
* PSA used as an eligibility criterion must be drawn within 42 days prior to injection number 1 and will be redrawn on Day 1 for use as a baseline value.

Exclusion Criteria:

* Candidates for salvage radiation therapy unless the patient refuses.
* Active or unresolved clinically significant infection.
* Parenteral antibiotics <7 days prior to initiation of treatment.
* Evidence of prior or current CNS metastases. Specific imaging is not necessary in the absence of signs or symptoms.
* Co-morbid medical conditions which would result in a life expectancy (participation) of less than 1 year.
* Patients with compromised immune systems; congenital, acquired, or drug-induced (immunosuppressive agents) will be excluded from the study. Use of prednisone at doses higher than 10 mg daily (or equipotent steroid doses) for more than 7 days within the last 3 months is not allowed.
* No-pre-existing malignancies that required treatment within the past 5 years except for basal or squamous cell cancers of the skin.
* Prior systemic therapies for prostate cancer not allowed (hormonal therapy, including but not limited to LHRH agonists, antiandrogens, ketoconazole or chemotherapy - mitoxantrone/taxanes/estramustine, etc.) except when patients stopped hormone therapy two or more years prior to enrollment and currently have normal testosterone levels; patients in Arm B, undergoing androgen depletion therapy during the vaccination will be eligible.
* Prior participation in any vaccine studies for non-infectious diseases.
* The inability to understand the language and the clinical protocol.
* Allergy or religious objection to pork products; Gelfoam is produced from pork.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Lubaroff, PhD, Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elzey BD, Siemens DR, Ratliff TL, Lubaroff DM. Immunization with type 5 adenovirus recombinant for a tumor antigen in combination with recombinant canarypox virus (ALVAC) cytokine gene delivery induces destruction of established prostate tumors. Int J Cancer. 2001 Dec 15;94(6):842-9. doi: 10.1002/ijc.1556. PMID 11745487
- [Background] Lubaroff DM, Konety B, Link BK, Ratliff TL, Madsen T, Shannon M, Ecklund D, Williams RD. Clinical protocol: phase I study of an adenovirus/prostate-specific antigen vaccine in men with metastatic prostate cancer. Hum Gene Ther. 2006 Feb;17(2):220-9. doi: 10.1089/hum.2006.17.220. No abstract available. PMID 16454655

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccine | Adenovirus/PSA Vaccine
Started | 25 | 25
Completed | 20 | 20
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccine | Adenovirus/PSA Vaccine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: years] | 71 [51 to 87] | 69 [58 to 84] | 70 [51 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 25 | 23 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop a Strong or Modest Anti-PSA Immune Response
Description: Anti-immunologic response is defined as an increase of >200% above pre-immunization levels of anti-PSA T cells as measured by ELISPOT analysis
Time Frame: 18 months
Population: 21 evaluable participants analyzed on Arm A and included in analysis of outcome measure one. 1 participant was lost to long-term follow-up for outcome measure three.
Measure: Number; unit: participants
Groups:
- Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccin: On Arm B, subjects will be started on androgen deprivation therapy (ADT) 14 days prior to beginning the vaccinations.
  Adenovirus/PSA Vaccine: 1x10E8pfu in Gelfoam subcutaneously on day 0, 30, 60
Arm/Group | Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccin | Adenovirus/PSA Vaccine
Number analyzed (Participants) | 20 | 21
participants
  Stong response | 12 | 14
  Modest response | 6 | 3

2. Secondary Outcome: Number of Participants With Stable, Decreased, or Increased PSA Doubling Times (PSADT)
Description: To evaluate the increase, decrease, or stable response rates (PSA responses and changes in PSADT) of the Ad/PSA vaccine using a prime-boost immunization strategy. PSADT will be calculated based on the MSKCC online calculator.
Time Frame: 18 months
Population: PSA levels and doubling times could not be analyzed for participants in Arm B due to the fact that their ADT reduces serum PSA.
Measure: Number; unit: participants
Arm/Group | Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccine | Adenovirus/PSA Vaccine
Number analyzed (Participants) | 0 | 19
participants
  Decreased PSADT |  | 4
  Stable PSADT |  | 2
  Increased PSADT/PSA decline |  | 13

3. Secondary Outcome: Number of Participants Alive and Deceased Following Treatment
Description: To evaluate survival in evaluable patients receiving the Ad/PSA vaccine, as measured by 2-year, 5-year, 10-year, and overall survival (OS)
Time Frame: Every 6 months, up to 14 years
Population: 5 participants lost to follow-up in Arm A, 5 participants lost to follow-up in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccine | Adenovirus/PSA Vaccine
Number analyzed (Participants) | 20 | 20
Participants
  2-year survival: Alive | 20 | 20
  2-year survival: Deceased | 0 | 0
  5-year survival: Alive | 19 | 20
  5-year survival: Deceased | 1 | 0
  10-year survival: Alive | 14 | 11
  10-year survival: Deceased | 6 | 9
  Overall survival: Alive | 3 | 10
  Overall survival: Deceased | 17 | 10

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was collected and assessed every 6 months via phone and then via medial record review during long-term follow-up, up to 14 years, AEs collected and recorded at least 4 weeks (30 days) after the last exposure to the study drug (up to day 90).
Groups:
- Adenovirus/PSA Vaccin: On Arm A, subjects can begin the three vaccinations immediately.
  Adenovirus/PSA Vaccine: 1x10E8pfu in Gelfoam subcutaneously on day 0, 30, 60
Arm/Group | Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccine | Adenovirus/PSA Vaccin
All-Cause Mortality (participants affected / at risk) | 17/25 | 10/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 15/25 | 18/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Androgen Deprivation Therapy (ADT) + Adenovirus/PSA Vaccine (N=25) | Adenovirus/PSA Vaccin (N=25)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Increase voiding frequency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Facial flushing (Vascular disorders) | 1 (1) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain, GI; oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site reaction (Investigations) | 1 (1) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection, bug bites on skin (Infections and infestations) | 0 (0) | 1 (1)
Common cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sleeplessness (General disorders) | 1 (1) | 1 (1)
Hypertension (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Elevated leukocyte esterase (Renal and urinary disorders) | 0 (0) | 1 (1)
Tooth pain/extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Upper airway infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Drainage of cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Decreased libido (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Hot flashes (General disorders) | 11 (11) | 0 (0)
Increased urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Increased urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Increased erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flu (General disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated ALT (Investigations) | 1 (1) | 0 (0)
Elevated AST (Investigations) | 1 (1) | 0 (0)
Leg cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell cancer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic, other (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated LDH (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Eye hemorrhage (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-01-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT00583752/Prot_SAP_000.pdf
  • Informed Consent Form (2013-12-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT00583752/ICF_001.pdf